CLINICAL TRIAL: NCT00996320
Title: Effect of Reducing ICU Interns' Work Hours on Sleep, Intern Well-Being, and Medical Errors
Brief Title: Work Hour Reductions, Medical Errors, and Intern Well-Being at Providence St. Vincent Medical Center Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence St. Vincent Department of Medicine (Unknown); Providence Center for Outcomes Research and Education (Unknown)
Responsible Party: Michelle Schoepflin Sanders MD, Providence St. Vincent Department of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 08-74B
Record Dates: First submitted 2009-08-28; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Sleep Deprivation; Depression
Keywords: Internship and Residency; Medical Errors; Burnout, Professional; Burnout; Depression; Actigraphy; Personnel Staffing and Scheduling; Sleep Deprivation; Workload; Humans; Adult; Male; Female; Intensive Care Units; Prospective Studies; Crossover Studies; Work Schedule Tolerance; Disorders of Excessive Somnolence; Guideline Adherence; Internal Medicine Education
MeSH Terms: conditions — Sleep Deprivation; Depression; Burnout, Professional; Burnout, Psychological; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Schedule (Experimental): Interns on the intervention schedule work the a modified ICU schedule averaging about 60 hours per week over 4 weeks, with maximum scheduled shift length 16 hours.
  Interventions: Other: Reduced work hour schedule
- Traditional Schedule (No Intervention): Interns on the traditional schedule work the usual ICU schedule averaging about 80 hours per week over 4 weeks, with maximum shift length 30 hours.

INTERVENTIONS:
Other: Reduced work hour schedule — Interns on the intervention schedule work an average of 60 hours per week over 4 weeks, with maximum shift length 16 hours.
  Arms: Intervention Schedule

SUMMARY:
The purpose of this study is to determine whether reducing intern work hours and eliminating extended shifts in the intensive care unit will reduce prescribing errors and improve intern well-being.

DETAILED DESCRIPTION:
Each intern enrolled will complete three 4-week rotations in the intensive care unit (ICU) at Providence St. Vincent Medical Center. Each intern will complete at least one traditional schedule and one intervention schedule. The traditional schedule consists of an 80-hour work week with overnight call every third night. The longest shift on the traditional schedule is 30 hours. The intervention schedule consists of a 60-hour work week which eliminates overnight call by assigning a variety of shifts ranging from 8 to 16 hours in length.

ELIGIBILITY:
Inclusion Criteria:

* Interns rotating at Providence St. Vincent Medical Center ICU

Exclusion Criteria:

* Diagnosis of narcolepsy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Multiple Sleep Latency Test | Measured once a month for each intern while on ICU rotation, at least 14 days into the scheduled 28 day cycle

SECONDARY OUTCOMES:
Hours slept per night measured by actigraphy | Daily
Pharmaceutical order error rate | Daily
Burnout measured by Maslach Burnout Inventory | Measured once per month for each intern while on ICU rotation, at least 14 days into the 28 day rotation
Beck Depression Inventory, Second Edition (BDI-II) | Measured once per month for each intern while on ICU rotation, at least 14 days into the 28 day rotation
Hours worked per shift on the traditional and intervention schedules | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Schoepflin Sanders, MD, Principal Investigator — Providence St. Vincent Medical Center
Locations (1):
- Providence St. Vincent Medical Center Intensive Care Unit, Portland, Oregon, United States